CLINICAL TRIAL: NCT01009567
Title: Compare the Efficacy of Human Albumin With Cabergoline to Prevent of Ovarian Hyper Stimulation in ART Program
Brief Title: Compare the Efficacy of Human Albumin With Cabergoline to Prevent Ovarian Hyper Stimulation in Assisted Reproductive Technology (ART) Program
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Royan-Emb-004
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2009-11

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: OHSS
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator): Receive human albumin 20% infusion
  Interventions: Drug: Control
- Cabergoline (Experimental): Receive cabergoline tablet (0/5 mg) daily until 6 days after oocytes retrieval
  Interventions: Drug: Cabergoline

INTERVENTIONS:
Drug: Cabergoline — Receive cabergoline tablet (0/5 mg) daily until 6 days after oocytes retrieval
  Other Names: B
  Arms: Cabergoline
Drug: Control — Receive human albumin 20% infusion
  Other Names: A
  Arms: Control

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of cabergoline in prevention of ovarian hyperstimulation syndrome versus albumin in ART program.

DETAILED DESCRIPTION:
Ovarian hyperstimulation syndrome (OHSS) is a iatrogenic potentially life threatening complication of assisted reproduction technologies due to gonadotropin and human chorionic gonadotropin administration. Its severe form has been reported in 1-10% of in vitro fertilization cycles.

Different strategies have been proposed for the prevention of OHSS in high-risk patients, but these approaches do not offer complete protection against the development of ovarian hyperstimulation syndrome (OHSS). Among the selected preventive methods, discontinuing (coasting) gonadotropin therapy and i.v. albumin were by far the most popular choices. Several previous studies have shown that cabergoline is a safe drug, both for mother and conceptus, for the treatment of macroadenoma hyperprolactinemia. We think that this kind of therapy may be safe both for mother and conceptus (as previously shown by several studies on dopamine agonists treatment of hyperprolactinemia during pregnancy), easier, cheaper and probably, more effective than previous OHSS treatments (albumin, steroids, dopamine). There is an urgent need to test cabergoline efficacy in OHSS prevention in high risk patients with a large multicenter study.

The proposal of This study approved by our institutional review boards and institution's ethical committee, and all Participants will sign a written consent before enter to study. Patients entering the intracytoplasmic sperm injection (ICSI) / IVF program in Royan institute and infertility research center in Valieasr hospital in Iran. We use a downregulation protocol with a GnRH agonist (buserelin acetate) as a long protocol for ICSI/ IVF-ET. We evaluate patients for high risk factors of severe OHSS. The inclusion criterion was the collection of >20 oocytes during oocyte retrieval. They allocate by a series of computer-generated random into two groups after the oocytes retrieval. 30 minutes after oocytes retrieval patients in A Group , receive human albumin 20% infusion and in B group receive cabergoline tablet (0/5 mg) daily until 6 days after oocytes retrieval then women in all groups will informed about the signs and symptoms of OHSS and counsel to contact with our institute if OHSS develops. Patients will monitor routinely 6days after ET by ultrasonographic examination for ovarian size and for detection of ascites. Moderate to severe OHSS patients hospitalize and evaluate routinely by haematological and biochemical tests. OHSS patients diagnose and classify according to Golan et al 1989.we compare incidence of OHSS and severity of OHSS patients in two groups. Pregnant patients follow until the 12th gestational week.

ELIGIBILITY:
Inclusion Criteria:

* patients at risk of developing OHSS, defined by the development of 20-30 follicles larger than 12 mm in diameter and retrieval of more than 20 oocytes
* ovarian stimulation with long protocol

Exclusion Criteria:

* coasting cases

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Percentage and severity of OHSS in two groups | 6 days after embryos transfer (ET)

SECONDARY OUTCOMES:
Efficacy and safety of cabergoline and albumin | 6 days after embryos transfer (ET)

CONTACTS AND LOCATIONS:
Overall Officials: Eniseh Tehraninejad, MD, Study Director — Royan Institute; Ashraf Moini, MD, Study Director — Board scientific; Marzieh Shiva, MD, Principal Investigator — scientist
Locations (1):
- Endocrinology and Female Infertility Department, Reproductive Medicine Research Center, Royan institute, ACECR, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Tehraninejad ES, Hafezi M, Arabipoor A, Aziminekoo E, Chehrazi M, Bahmanabadi A. Comparison of cabergoline and intravenous albumin in the prevention of ovarian hyperstimulation syndrome: a randomized clinical trial. J Assist Reprod Genet. 2012 Mar;29(3):259-64. doi: 10.1007/s10815-011-9708-4. Epub 2012 Jan 10. PMID 22231013
- See also: Related Info — http://www.Royaninstitute.org